CLINICAL TRIAL: NCT05421377
Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Development of a Screening Set for Patients at Risk for Developing LLL
Brief Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Aim 2
Acronym: EvaLymph-Leg2
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Tessa De Vrieze, Post-doctoral research fellow and physiotherapist, PhD in Biomedical Sciences (Catholic University of Leuven) and Medical Sciences (University of Antwerp), KU Leuven
Other Study IDs: s66033-aim2
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Lower Limb Lymphedema
Keywords: screening; urogenital cancer; gynaecological cancer; skin cancer; lymph node dissection
MeSH Terms: conditions — Urogenital Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lymph node dissection for treatment of urogenital, gynaelogical or skin cancer: Patients with any type of skin melanoma (at the level of the lower limb), urogenital or gynaecological cancer scheduled for lymph node dissection
  Interventions: Diagnostic Test: clinical assessment

INTERVENTIONS:
Diagnostic Test: clinical assessment — screening of patients at risk for developing unilateral or bilateral lower limb lymphedema

SUMMARY:
Lymphedema is a chronic, debilitating disorder characterized by abnormal tissue swelling, adipose deposition and tissue fibrosis, resulting from disruption, blockage, or genetic abnormalities of the lymphatic system. Secondary lymphedema is an acquired lymphedema due to trauma, surgery, radiotherapy or infection among others resulting in a decreased transport capacity of the lymphatic system. This can be combined with an additional load on the lymphatic system due to obesity, venous hypertension or a wound, among others. Advances in oncologic treatment have led to an ever-increasing number of cancer survivors over time. As a result, morbidities related to this treatment (such as secondary lymphedema) are likely to increase too.

Risk factors for the development of LLL after treatment for (gynaecological) cancer are: pelvic and para-aortic lymphadenectomy, the number of pelvic lymph nodes removed, adjuvant radiotherapy, adjuvant chemotherapy, increasing BMI/ BMI ≥25 kg/m², lymphocyst formation, increasing age, increasing time since surgery and insufficient physical activity level.

To the investigators knowledge, no evidence exists regarding which (combination of) measuring methods are most sensitive to detect early lymphedema at the lower limbs after the treatment of cancer. Thresholds for identifying subclinical edema on one or both lower limbs are lacking.

Therefore the investigators want to develop a screening set for patients at risk for developing LLL. Which measurement method (and which criterion) shows the best diagnostic accuracy in screening patients at risk for LLL after cancer treatment? And: What is the added value of combining different measurement methods in terms of diagnostic accuracy?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of skin melanoma (at the level of the lower limb, at least cancer stage 3), gynecological cancer, uro-genital cancer that will receive surgery (sentinel lymph node biopsy and/or (para-aortic/inguinal/pelvic) lymph node dissection)

Exclusion Criteria:

* Pregnant participants
* Presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Presence of skin infections of wounds at the level of the lower limbs at the moment of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at risk for LLL (i.e. patients undergoing pelvic/inguinal/para-aortic lymph node dissection for uro-genital, gynaecological or skin cancer) will be included from pre-surgery up to 12 months post-surgery
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of reliable and clinical feasible measurement methods regarding the screening of patients at risk for developing unilateral or bilateral LLL | up to 12 months post-surgery
  Sensitivity of reliable and clinical feasible measurement methods (resulted from aim 1: NCT05269264) regarding the screening of patients at risk for developing unilateral or bilateral LLL at 6 weeks, 6, and 12 months post-surgery
Specificity of reliable and clinical feasible measurement methods regarding the screening of patients at risk for developing unilateral or bilateral LLL | up to 12 months post-surgery
  Specificity of reliable and clinical feasible measurement methods (resulted from aim 1: NCT05269264) regarding the screening of patients at risk for developing unilateral or bilateral LLL at 6 weeks, 6, and 12 months post-surgery
Diagnostic accuracy of reliable and clinical feasible measurement methods regarding the screening of patients at risk for developing unilateral or bilateral LLL | up to 12 months post-surgery
  Diagnostic accuracy of reliable and clinical feasible measurement methods (resulted from aim 1: NCT05269264) regarding the screening of patients at risk for developing unilateral or bilateral LLL at 6 weeks, 6, and 12 months post-surgery

SECONDARY OUTCOMES:
Prognostic value of 'baseline age' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Age (years) will be self-reported through interview.
Prognostic value of 'baseline age' for the development of bilateral lower limb lymphoedema at 12 months post-surgery. | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Age (years) will be self-reported through interview.
Prognostic value of ' Baseline physical activity level' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Baseline physical activity level : will be assessed with the International Physical Activity Questionnaire (IPAQ).
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Prognostic value of ' Baseline physical activity level' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Baseline physical activity level : will be assessed with the International Physical Activity Questionnaire (IPAQ).
  The IPAQ is a 27-item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Prognostic value of ' Baseline educational level' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Educational level: will be self-reported through interview.
Prognostic value of ' Baseline educational level' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Educational level: will be self-reported through interview.
Prognostic value of ' Baseline BMI' for the development of bilateral lower limb lymphoedema at 6 weeks post- surgery | 6 weeks post- surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= baseline Body Mass Index
Prognostic value of ' Baseline BMI' for the development of bilateral lower limb lymphoedema at 12 months post- surgery | 12 months post- surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= baseline Body Mass Index
Prognostic value of ' Baseline comorbidities' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= baseline comorbidities
  Comorbidities will be reported through a self-developed co-morbidity questionnaire, based on IDEWE questionnaire.
Prognostic value of ' Baseline comorbidities' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= baseline comorbidities
  Comorbidities will be reported through a self-developed co-morbidity questionnaire, based on IDEWE questionnaire.
Prognostic value of 'Type of cancer' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Type of cancer Information regarding the type of cancer is collected by exploring the patient's medical file.
Prognostic value of 'Type of cancer' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Type of cancer Information regarding the type of cancer is collected by exploring the patient's medical file.
Prognostic value of 'Tumor stage' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | at 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Tumor stage
  Information regarding the tumor stage of is collected by exploring the patient's medical file.
Prognostic value of 'Tumor stage' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Tumor stage
  Information regarding the tumor stage of is collected by exploring the patient's medical file.
Prognostic value of 'Lymph node stage' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Lymph node stage
  Information regarding the lymph node stage of is collected by exploring the patient's medical file.
Prognostic value of 'Lymph node stage' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable= Lymph node stage
  Information regarding the lymph node stage of is collected by exploring the patient's medical file.
Prognostic value of 'Number of positive lymph nodes' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable=Number of positive lymph nodes: is collected through the patient's medical file.
Prognostic value of 'Number of positive lymph nodes' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Dependent variable = presence of lower limb lymphoedema Independent variable=Number of positive lymph nodes: is collected through the patient's medical file.
Prognostic value of 'Postoperative complications' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Information regarding the complications related to the surgery as well as adjuvant therapies is collected. Surgical complications will be assessed according to the Clavien-Dindo Classification of Surgical Complications.
Prognostic value of 'Postoperative complications' for the development of lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Information regarding the complications related to the surgery as well as adjuvant therapies is collected. Surgical complications will be assessed according to the Clavien-Dindo Classification of Surgical Complications.
Prognostic value of 'Type of lymph node dissection' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
  Type of lymph node dissection: Limited- Standard- Extended- Super extended
Prognostic value of 'Type of lymph node dissection' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
  Type of lymph node dissection: Limited- Standard- Extended- Super extended
Prognostic value of 'Number of lymph nodes removed' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
Prognostic value of 'Number of lymph nodes removed' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Cancer treatment characteristics are collected (i.e. type of surgery, type of lymph node dissection, number of lymph nodes removed, presence of postoperative drain, number of positive lymph nodes, adjuvant therapies; by exploring the patient's medical file.
Prognostic value of 'Adjuvant Radiotherapy' for the development of bilateral lower limb lymphoedema at 6 weeks post-surgery | 6 weeks post-surgery
  Cancer treatment characteristics , including adjuvant radiotherapy are collected; by exploring the patient's medical file.
Prognostic value of 'Adjuvant Radiotherapy' for the development of bilateral lower limb lymphoedema at 12 months post-surgery | 12 months post-surgery
  Cancer treatment characteristics , including adjuvant radiotherapy are collected; by exploring the patient's medical file.
Incidence rate of unilateral and bilateral LLL at 6 weeks post-surgery | 6 weeks post-surgery
  Calculation of the proportion of patients with leg (or foot) lymphedema, defined as 5.0% or more increase of the leg (or foot) volume in each leg (or foot), at a certain time point, compared to the volumes at baseline; OR patients with a score of at least 5 out of 52 on the detect-OL questionnaire in case it is clearly indicated whether symptoms are present in one or both legs (in order to be able to categorize patients to the "unilateral LLL" or "bilateral LLL" group).
  Additionally, the proportion of presence of LLL in patients having received a lymph node dissection due to gynaecological cancer vs. due to urogenital cancer vs. due to skin melanoma will be compared. The distribution of LLL (unilateral vs. bilateral, regions of the lower limb) will be encountered and compared.
Incidence rate of unilateral and bilateral LLL at 6 months post-surgery | 6 months post-surgery
  Calculation of the proportion of patients with leg (or foot) lymphedema, defined as 5.0% or more increase of the leg (or foot) volume in each leg (or foot), at a certain time point, compared to the volumes at baseline; OR patients with a score of at least 5 out of 52 on the detect-OL questionnaire in case it is clearly indicated whether symptoms are present in one or both legs (in order to be able to categorize patients to the "unilateral LLL" or "bilateral LLL" group).
  Additionally, the proportion of presence of LLL in patients having received a lymph node dissection due to gynaecological cancer vs. due to urogenital cancer vs. due to skin melanoma will be compared. The distribution of LLL (unilateral vs. bilateral, regions of the lower limb) will be encountered and compared.
Incidence rate of unilateral and bilateral LLL at 12 months post-surgery | 12 months post-surgery
  Calculation of the proportion of patients with leg (or foot) lymphedema, defined as 5.0% or more increase of the leg (or foot) volume in each leg (or foot), at a certain time point, compared to the volumes at baseline; OR patients with a score of at least 5 out of 52 on the detect-OL questionnaire in case it is clearly indicated whether symptoms are present in one or both legs (in order to be able to categorize patients to the "unilateral LLL" or "bilateral LLL" group).
  Additionally, the proportion of presence of LLL in patients having received a lymph node dissection due to gynaecological cancer vs. due to urogenital cancer vs. due to skin melanoma will be compared. The distribution of LLL (unilateral vs. bilateral, regions of the lower limb) will be encountered and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa De Vrieze, Dr., Principal Investigator — KU Leuven
Locations (1):
- University Hospitals of Leuven, Leuven, Belgium